CLINICAL TRIAL: NCT01872403
Title: Neoadjuvant Chemotherapy of Nanoparticle Albumin-bound Paclitaxel/Carboplatin vs. Paclitaxel /Carboplatin in Stage Ⅱ B and IIIA Squamous Cell Carcinoma of the Lung: Parallel Control and Single Center
Brief Title: Neoadjuvant Chemotherapy of Nanoparticle Albumin-bound Paclitaxel/Carboplatin vs. Paclitaxel /Carboplatin in Stage Ⅱ B and IIIA Squamous Cell Carcinoma of the Lung
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, The First Affiliated Hospital of Guangzhou Medical University, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAH20120906; FAHGuangzhou011 (Registry Identifier: FAHGuangzhou)
Record Dates: First submitted 2013-05-15; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Squamous Cell Carcinoma of the lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Taxes; Carboplatin; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nanoparticle albumin-bound paclitaxel (Experimental): Neoadjuvant chemotherapy of nanoparticle albumin-bound paclitaxel/carboplatin in stage Ⅱ B and IIIA squamous cell carcinoma of the lung
  Interventions: Drug: nanoparticle albumin-bound paclitaxel/carboplatin

INTERVENTIONS:
Drug: nanoparticle albumin-bound paclitaxel/carboplatin — Neoadjuvant chemotherapy of nanoparticle albumin-bound paclitaxel/carboplatin vs. paclitaxel /carboplatin in stage Ⅱ B and IIIA squamous cell carcinoma of the lung:
  Other Names: paclitaxel /carboplatin

SUMMARY:
Albumin-bound paclitaxel plus carboplatin regimen in advanced NSCLC especially in lung squamous cell carcinoma has a better tumor response rate and safety, therefore.The main purpose of this study is to observe the safety and efficacy of albumin-bound paclitaxel / carboplatin in the treatment of lung squamous cell carcinoma of stage IIB and IIIA.

DETAILED DESCRIPTION:
Albumin-bound paclitaxel plus carboplatin regimen in advanced NSCLC especially in lung squamous cell carcinoma has a better tumor response rate and safety, therefore, this program is applied to neoadjuvant therapy, may obtain better tumor pathological remission rate, improve the operation resection rate, thus improve the prognosis.The main purpose of this study is to observe the safety and efficacy of albumin-bound paclitaxel / carboplatin in the treatment of lung squamous cell carcinoma of stage IIB and IIIA.

ELIGIBILITY:
Inclusion Criteria:

1.Histological or cytological diagnosis of lung squamous cell carcinoma of stage IIB and IIIA.

2.18 years or older 3.ECOG Performance Status no more than 2; 4.Appraisable disease, the presence of at least three lesions if longest diameter <10 mm by brain MRI; 5.Haemoglobin 10.0 g/dl, Absolute neutrophil count (ANC) 1.5 x 10E9/L, platelets 100 x 10E9/L; 6.Total bilirubin 1.5 x upper limit of normal (ULN); 7.ALT and AST < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases; 8.Creatinine clearance 60ml/min (calculated according to Cockcroft-gault formula).

Exclusion Criteria:

1. Any systemic anticancer treatment for NSCLC
2. Local radiotherapy for NSCLC.
3. In this study within five years prior to the start of treatment with other than NSCLC patients with other cancers.
4. Any instability in systemic disease, including: active infection, absence of control hypertension, unstable angina, begins in the last 3 months of angina pectoris, congestive heart failure
5. HIV infection;
6. Allergic to paclitaxel or Platinum;
7. mixed with adenocarcinoma, small cell lung cancer;
8. Pregnant or lactating women;
9. Other researchers believe that does not fit into the group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Tumor ORR and Number of Adverse Events | From date of randomization until the date of progression, assessed up to 2 months

SECONDARY OUTCOMES:
PFS | From date of surgery until the date of first documented progression, assessed up to 30 months

OTHER OUTCOMES:
The rate of pathology down-stage of lymph nodes | 1 day (the date of surgery)

CONTACTS AND LOCATIONS:
Overall Officials: jianxing he, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China